CLINICAL TRIAL: NCT05429060
Title: A Prospective Assessment of Surgical Treatments in Hemorrhoidal Disease: Real-life Practice and Early Outcome in Terms of Patient-reported Symptoms and Quality of Life
Brief Title: A Prospective Evaluation of Hemorrhoidal Surgery Outcome in Istanbul
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-10840098-772.02-109
Record Dates: First submitted 2022-05-11; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Hemorrhoids; Quality of Life; Complication of Treatment; Indication, Unlabeled
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hemorrhoidal surgery — All surgical interventions under general or local anesthesia, either in the office or operation room, including any type of injection, excision, ligation, ablation, mucopexy and suturation.

SUMMARY:
This study aims to evaluate the effect of surgical treatments on the quality of life in hemorrhoidal disease. All available treatment methods will be included in this 1-year cohort which is going to collect data from a big metropol.

ELIGIBILITY:
Inclusion Criteria:

* Surgical interventions under local and/or general anesthesia
* Elective or emergency interventions (including thrombectomy)
* Surgical interventions in operation room or office
* Any kind of excision, sclerotherapy, ligation, suturation, ablation, mucopexy

Exclusion Criteria:

* Any accompanying perianal disease (anal fistula, anal fissure, perianal abscess, anal condyloma extending into the anal canal)
* Previous surgery for hemorrhoids (any intervention other than medical treatment)
* Previous perianal surgery (internal sphincterotomy, fistula surgery)
* Pelvic and/or perineal radiotherapy
* Previous obstetric or perianal injury and/or sphincter repair
* Previous rectal surgery (distal colectomy for benign or malignant etiology)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults who underwent any interventional treatment other than medical therapy under local and/or general anesthesia will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Short Health Scale-HD score at 1 year after hemorrhoidal surgery | 1 year
  Changes in quality of life from baseline at 1 year in terms of Short Health Scale (SHS) specific to hemorrhoidal disease (HD) will be reported for each surgical treatment. The SHS-HD scores will be recorded preoperatively, at 1 week, 6 weeks, and 12 months.
Hemorrhoidal Disease Symptom Score at 1 year after hemorrhoidal surgery | 1 year
  Changes in symptoms from baseline at 1 year will be reported for each surgical treatment. Hemorrhoidal Disease Symptom Score (HDSS) described by Nyström based on 5 cardinal symptoms (pain, itching, bleeding, soiling, and prolapse) will be recorded preoperatively, at 1 week, 6 weeks, and 12 months.

SECONDARY OUTCOMES:
Recurrence | 1 year
  Determining recurrence rate at 1 year for each treatment. Relapse of patient-reported symptoms (pain, itching, bleeding, soiling, and prolapse) will be recorded at 1 year.
Complications | 1 year
  Determining early and late complications for each treatment. Early complications (abscess, urinary retention) will be assessed at 6 weeks. Late complications (incontinence, anal stenosis) will be assessed at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Cigdem Arslan, MD, Study Director — Medipol University
Locations (1):
- Medipol University Bahcelievler Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kement M, Tekin A, Baysal H, Tosun S, Alimoglu O, Sucullu I, Civil O, Sakoglu N, Arslan NC, Tatar C, Nayci AE, Ari A, Cakir E, Kaya R, Turan I, Gulsen T, Meric S, Yavuz E, Bugdayci N, Hamad FM, Leventoglu S, Kozan R, Akpinar O, Yanar H, Yanar F, Kucuk HF, Karahan M, Kaya S, Adiguzel NC, Onder T, Abci I, Aydin AZ, Ozkan OF, Kiziltoprak N, Ozcan B, Orhan A, Canturk AO, Tan M, Bilgin Y, Cok H, Cezit A, Fersahoglu MM, Oncel M. Patient-reported outcomes after hemorrhoid surgery: early results from a prospective, nationwide, real-world, cohort study on diverse approaches. Ann Coloproctol. 2025 Dec;41(6):573-585. doi: 10.3393/ac.2025.00710.0101. Epub 2025 Dec 30. PMID 41486915